CLINICAL TRIAL: NCT01317797
Title: A Phase Ib Double-blind, Placebo-controlled, Randomized, Dose-escalating Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Efficacy of Repeated Subcutaneous Injections of MT203 in Patients With Mild to Moderate Rheumatoid Arthritis on Treatment With Methotrexate
Brief Title: A Trial to Evaluate the Safety and Tolerability of Namilumab (MT203) in Patients With Mild to Moderate Rheumatoid Arthritis
Acronym: PRIORA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M1-1188-002-EM; 2010-018502-36 (EudraCT Number); U1111-1137-3923 (Registry Identifier: WHO); NL33507.058.10 (Registry Identifier: CCMO)
Record Dates: First submitted 2011-02-18; First posted 2011-03-17 (Estimated); Results first posted 2015-08-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; MT203; Human IgG1 monoclonal antibody; GM-CSF monoclonal antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — namilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Namilumab 150 mg (Experimental): Namilumab (MT203) 150 mg (low dose), subcutaneous (SC) injection, on Days 1, 15 and 29.
  Interventions: Drug: namilumab (MT203)
- Namilumab 300 mg (Experimental): Namilumab (MT203) 300 mg (high dose), SC injection, on Days 1, 15 and 29.
  Interventions: Drug: namilumab (MT203)
- Placebo (Placebo Comparator): Namilumab-matching placebo, SC injection, on Days 1, 15 and 29.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: namilumab (MT203) — administered three times, subcutaneous in the abdomen
  Arms: Namilumab 150 mg; Namilumab 300 mg
Drug: Placebo — administered three times, subcutaneous in the abdomen
  Arms: Placebo

SUMMARY:
The purpose of this trial is primarily to investigate the safety and tolerability of repeated subcutaneous injections of MT203 in patients with mild to moderate rheumatoid arthritis. Furthermore, the amount of MT203 in the blood will be measured and it will be investigated how the body responds to MT203 treatment and if MT203 is effective in the treatment of rheumatoid arthritis.

DETAILED DESCRIPTION:
The trial medication will be administered at 2 dose levels as subcutaneous injections. Each patient will receive three injections in total. The trial duration consists of a screening period (28 - 2 days prior to the first injection) and a treatment and observation period (4 months). The trial requires approximately 20 visits at the study site.

ELIGIBILITY:
Inclusion Criteria:

1. Out-patients with active rheumatoid arthritis (RA), according to the ACR 1987 revised criteria, with low to moderate disease activity (DAS28-ESR ≥ 2.6 and ≤ 5.1)
2. Patients must be on stable doses of methotrexate (MTX) ≥ 7.5 and ≤ 25 mg/week for at least 12 weeks before the first injection, with appropriate folic acid supplementation
3. Age ≥ 18 years at Screening
4. Body weight at least 50 kg at Screening; BMI: ≥ 18.0 and ≤ 30.0 kg/m2 at Screening
5. Negative tuberculosis test at Screening
6. Heterosexually active male and female patients of childbearing potential are obliged to follow whatever contraceptive and / or breastfeeding restrictions may be required for their concomitant medication(s), including methotrexate.

In addition, heterosexually active male and female patients of childbearing potential are required to use effective double-method contraception (one hormonal contraceptive or intrauterine device and one other additional contraceptive method) for 1 month before the first administration of the IMP, during the course of the trial, and for 6 month after the last injection of MT203.

No special requirements are made for female patients proven to be post-menopausal (at least 2 years after last menstrual period and FSH ≥ 40IU/L), surgically sterilized or hysterectomized. Likewise no special requirements for heterosexually active male who are surgical sterilized.

Pregnant or lactating female patients have to be excluded.

Exclusion Criteria:

1. Participation in another clinical trial or previous dosing in this trial
2. Use of specified medications within certain timeframes or use of certain comedications
3. History or presence of specified diseases
4. Drug abuse
5. Certain laboratory parameters outside a specified range
6. Donation of blood
7. Relevant decrease in lung function
8. Infections, frequent or chronic infections, herpes zoster
9. Females: positive pregnancy test
10. Presence of history of tuberculosis
11. History of malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Nycomed Investigational Site, Sofia, Bulgaria
- Nycomed Investigational Site, Leids, Netherlands

REFERENCES:
- [Derived] Huizinga TW, Batalov A, Stoilov R, Lloyd E, Wagner T, Saurigny D, Souberbielle B, Esfandiari E. Phase 1b randomized, double-blind study of namilumab, an anti-granulocyte macrophage colony-stimulating factor monoclonal antibody, in mild-to-moderate rheumatoid arthritis. Arthritis Res Ther. 2017 Mar 9;19(1):53. doi: 10.1186/s13075-017-1267-3. PMID 28274253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 10 investigative sites in Bulgaria, Netherlands and Spain from 09 March 2011 to 08 August 2013.
Pre-assignment Details: Participants with a diagnosis of mild or moderate rheumatoid arthritis were enrolled into 1 of 3 treatment groups namilumab (MT203) 150mg, namilumab 300 mg or placebo.
Period: Overall Study
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Started | 8 | 7 | 9
Completed | 8 | 6 | 8
Not Completed | 0 | 1 | 1
Not completed — Other | 0 | 1 | 0
Not completed — Withdrawal of Patient | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo | Total
Number analyzed (Participants) | 8 | 7 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (6.95) | 56.6 (15.28) | 53.4 (11.05) | 55.9 (11.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 17
  Male | 3 | 1 | 3 | 7
Race/Ethnicity, Customized [Number; unit: participants]
  White | 7 | 7 | 9 | 23
  Black | 1 | 0 | 0 | 1
Height [Mean (Standard Deviation); unit: cm] | 166.21 (8.605) | 168.57 (6.321) | 168.44 (5.126) | 167.74 (6.581)
Weight [Mean (Standard Deviation); unit: kg] | 68.13 (7.140) | 80.44 (7.305) | 77.80 (8.617) | 75.35 (9.147)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 24.69 (2.471) | 28.30 (1.778) | 27.37 (2.246) | 26.75 (2.607)
Disease Activity Score 28-Erythrocyte Sedimentation Rate (DAS28-ESR) Score [Mean (Standard Deviation); unit: score on a scale] — The DAS28-ESR is expressed on a unit on a scale with the minimum score=0 (best) to maximum score=10 (worst).
  score on a scale | 4.70 (0.542) | 4.66 (0.544) | 4.60 (0.512) | 4.65 (0.510)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Clinical Laboratory Results
Description: Blood was collected for Haematology, Chemistry and Coagulation. Urine was collected for Urinalysis. Alert values for laboratory results include the following: Aspartate aminotransferase (ASAT), alanine aminotransferase (ALAT), gamma-glutamyl-transpeptidase (GGT), alkaline phosphatase (AP), total bilirubin (TBil): > 3 times upper limit of normal (ULN). Creatinine and Glucose: > 2 times ULN. Potassium > 6.0 or < 3.0 mmol/L. Haemoglobin: Male < 8.0 ;Female < 7.0 g/dL. Erythrocytes :Male < 3.5 x 10^12/L or > 7 x 10^12/L;Female < 3.0 x 10^12/L or > 6.5 x 10^12/L. White Blood Cells (WBC): < 2.8 x10^9/L or > 16.0 x 10^9/L. Eosinophils > 20 % of cells in the WBC differential. Platelet Count < 75 x 10^9/L or 600 x 10^9/L. No alert values were identified for Coagulation or Urinalysis.
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants
  Haematology | 3 | 0 | 1
  Chemistry | 1 | 1 | 1
  Coagulation | 0 | 0 | 0
  Urine | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Findings
Description: Alert values for ECG were: Heart rate < 35 bpm or > 120 bpm, QTc acc. to Bazett (absolute value)> 500 ms or QTc acc. to Bazett (increase versus Baseline (pre-treatment).
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs included Systolic Blood Pressure (BP), Diastolic BP, body temperature, heart rate. Alert values were: BP systolic > 170 mmHg or < 85 mmHg, BP diastolic > 105 mmHg, Difference BP systolic vs. Baseline (pre-treatment) > 40 mmHg or Pulse rate < 35 bpm or > 120 beats per minute (bpm).
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants | 3 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Pulmonary Function Tests
Description: Pulmonary function was determined by forced expiratory volume in the first second (FEV1), forced vital capacity (FVC) and peak flow.
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Findings
Description: The physical examination included body system assessments: eyes, head and neck (including thyroid), ears, nose and throat, lymph nodes, cardiovascular, lungs, mammae, abdomen (liver, spleen), genitals, limbs, central and peripheral nervous system, musculoskeletal system, skin & nails, mucosae. The Investigator classified abnormal findings as either clinically significant or not clinically significant.
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants | 0 | 0 | 0

6. Primary Outcome: Number of Participants Reporting One or More Treatment Emergent Adverse Events
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants | 5 | 4 | 5

7. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MT203
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax
Time Frame: Day 1 and 29 (Pre-dose and 2 and 6 hours post-dose)
Measure: Median (Full Range); unit: days
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 7
days
  Day 1 | 4.98 [3.0 to 7.0] | 5.95 [4.0 to 8.2]
  Day 29 | 4.97 [0.1 to 8.0] | 6.00 [1.0 to 13.0]

8. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for MT203
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: Day 1 and 29 (Pre-dose and 2 and 6 hours post-dose)
Population: PK Analysis set included all 15 participants who were exposed to study drug for whom any PK parameters could be calculated. Method of Dispersion is the 68% range.
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 7
μg/mL
  Day 1 | 13.41 [9.988 to 18.02] | 18.76 [13.83 to 25.45]
  Day 29 | 27.14 [22.02 to 33.45] | 49.99 [40.36 to 61.91]

9. Secondary Outcome: AUC(0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for MT203
Description: AUC(0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC[0-tlqc]).
Time Frame: Day 1 and 29 (Pre-dose and 2 and 6 hours post-dose)
Population: as for outcome 8
Measure: Geometric Mean (Full Range); unit: day*μg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 7
day*μg/mL
  Day 1 | 144.9 [112.3 to 186.9] | 210.9 [151.8 to 292.9]
  Day 29 | 786.8 [666.9 to 928.3] | 1696 [1293 to 2225]

10. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for MT203
Description: AUC(0-inf) is measure of area under the curve over the dosing interval (tau) (AUC(0-tau]), where tau is the length of the dosing interval in this study).
Time Frame: Day 29 (Pre-dose and 2 and 6 hours post-dose)
Population: as for outcome 8
Measure: Geometric Mean (Full Range); unit: day*μg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 6
day*μg/mL | 832.8 [708.8 to 978.4] | 1861 [1374 to 2521]

11. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for MT203
Description: Area under the plasma concentration-time curve during a dosing interval, where tau is the length of the dosing interval.
Time Frame: Day 29 (Pre-dose and 2 and 6 hours post-dose)
Population: as for outcome 8
Measure: Geometric Mean (Full Range); unit: day*μg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 7
day*μg/mL | 318.5 [263.2 to 385.5] | 591.9 [473.3 to 740.3]

12. Secondary Outcome: Terminal Phase Elimination Half-life (T1/2) for MT203
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: Day 29 (Pre-dose and 2 and 6 hours post-dose)
Population: PK Analysis set included all 15 participants who were exposed to study drug for whom any PK parameters could be calculated.
Measure: Mean (Full Range); unit: days
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 6
days | 21.26 [13.7 to 34.6] | 23.68 [18.6 to 29.9]

13. Secondary Outcome: Ctrough: Maximum Observed Plasma Concentration Pre-Dose
Time Frame: Days 1, 15 and 29 Pre-dose
Population: as for outcome 8
Measure: Geometric Mean (Full Range); unit: μg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg
Number analyzed (Participants) | 8 | 7
μg/mL
  Day 1 | 9.232 [7.543 to 11.30] | 14.56 [11.33 to 18.72]
  Day 15 | 15.53 [13.03 to 18.50] | 27.28 [18.89 to 39.41]
  Day 29 | 20.27 [16.74 to 24.53] | 36.88 [31.85 to 42.70]

14. Secondary Outcome: Change From Baseline in Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) in Plasma
Description: MT203/GM-CSF complexes were analysed using a procedure that quantified GM-CSF after dissociation from the complex. The determined concentrations corresponded to the amount of total (free and complexed) GM-CSF in the plasma sample. A positive change from Baseline indicated improvement.
Time Frame: Baseline and Days 2, 4, 6, 8 15, 29, 30, 35, 43, 56, 71, 99, End of trial (EOT) Up to Day 118
Population: All randomized participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
pg/mL
  Day 2 (n=7, 7, 9) | 0.00 (0.000) | -0.86 (2.268) | 0.67 (2.000)
  Day 4 (n=6, 7, 9) | 3.00 (3.286) | 0.86 (4.140) | 0.00 (0.000)
  Day 6 (n=6, 7, 9) | 3.00 (3.286) | 2.57 (3.207) | 0.00 (0.000)
  Day 8 (n=6, 7, 9) | 7.78 (10.330) | 4.29 (2.928) | 0.00 (0.000)
  Day 15 (n=7, 7, 9) | 16.86 (8.825) | 8.61 (8.978) | 0.00 (0.000)
  Day 29 (n=7, 7, 8) | 31.59 (13.323) | 15.14 (6.690) | 0.00 (0.000)
  Day 30 (n=6, 7, 8) | 40.68 (24.908) | 22.11 (16.954) | 0.75 (2.121)
  Day 35 (n=7, 7, 7) | 33.29 (20.203) | 25.71 (16.261) | 0.00 (0.000)
  Day 43 (n=7, 7, 8) | 40.04 (18.838) | 28.10 (15.013) | 0.00 (0.000)
  Day 56 (n=7, 6, 8) | 38.34 (20.330) | 32.32 (14.337) | 0.75 (2.121)
  Day 71 (n=5, 6, 8) | 31.48 (21.759) | 35.02 (12.402) | 0.75 (2.121)
  Day 99 (n=7, 6, 7) | 9.11 (11.113) | 23.77 (8.881) | 0.00 (0.000)
  EOT (n=7, 6, 9) | 3.87 (7.919) | 17.38 (10.745) | 0.67 (2.000)

15. Secondary Outcome: Change From Baseline in MT203/GM-CSF Complexes in Plasma
Description: as for outcome 14
Time Frame: Baseline and Days 2, 4, 6, 8 15, 29, 30, 35, 43, 56, 71, 99, EOT Up to Day 118
Population: All randomized participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
pg/mL
  Day 2 (n=8, 7, 9) | 30.9 (63.92) | 12.7 (16.25) | -0.2 (0.67)
  Day 4 (n=8, 7, 9) | 210.6 (183.16) | 186.1 (100.15) | -0.6 (1.67)
  Day 6 (n=8, 7, 9) | 381.6 (152.52) | 334.6 (89.19) | -1.3 (4.00)
  Day 8 (n=8, 7, 9) | 448.0 (110.76) | 534.1 (80.58) | -1.3 (4.00)
  Day 15 (n=8, 7, 9) | 1021.0 (353.03) | 1055.0 (124.65) | -3.9 (11.67)
  Day 29 (n=8, 7, 8) | 1566.9 (391.80) | 1805.4 (150.43) | -4.4 (12.37)
  Day 30 (n=8, 7, 8) | 1653.5 (498.31) | 1834.9 (178.71) | -4.4 (12.37)
  Day 35 (n=8, 7, 8) | 1796.9 (560.58) | 2052.9 (294.95) | -4.4 (12.37)
  Day 43 (n=8, 7, 8) | 2213.0 (744.37) | 2290.6 (282.35) | -4.4 (12.37)
  Day 56 (n=8, 6, 8) | 2009.0 (614.92) | 2457.2 (466.01) | -4.4 (12.37)
  Day 71 (n=8, 6, 8) | 1299.6 (313.20) | 2312.2 (492.50) | -4.4 (12.37)
  Day 99 (n=8, 6, 8) | 462.6 (275.40) | 1753.5 (351.34) | -4.4 (12.37)
  EOT (n=8, 6, 9) | 310.4 (144.03) | 1310.8 (460.45) | -3.9 (11.67)

16. Secondary Outcome: Number of Participants With Anti-MT203 Antibodies
Description: Serum samples were tested for the presence of anti-MT203 antibodies by a bridging Electro-chemi-luminescent assay (ECL-assay).
Time Frame: From Day 1 Up to Day 118
Population: Safety population included all randomized participants who received study drug.
Measure: Number; unit: participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
participants | 0 | 0 | 0

17. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR 20) Response
Description: ACR20 response is defined as a ≥ 20% improvement (reduction) compared with baseline for both total joint count-68 joints (TJC68) and swollen joint count-66 joints (SJC66), as well as for three of the additional five ACR core set variables: Patient's Assessment of Pain over the previous 24 hours: using a Visual Analog Scale (VAS) left end of the line 0=no pain to right end of the line 100=unbearable pain; Patient's Global Assessment of Disease Activity and Physician's Global Assessment of Disease Activity over the previous 24 hours using a VAS where left end of the line 0=no disease activity to right end of the line 100=maximum disease activity; Health Assessment Questionnaire: 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities, 0=without difficulty to 3=unable to do; and acute-phase reactant Erythrocyte Sedimentation Rate.
Time Frame: Baseline and Days 13,27,43,56,71,99 and EOT Up to Day 118
Population: All randomized participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
percentage of participants
  Day 13 | 50.0 | 14.3 | 11.1
  Day 27 | 50.0 | 57.1 | 33.3
  Day 43 | 37.5 | 71.4 | 44.4
  Day 56 | 50.0 | 57.1 | 55.6
  Day 71 | 62.5 | 57.1 | 44.4
  Day 99 | 50.0 | 42.9 | 44.4
  EOT | 37.5 | 57.1 | 44.4

18. Secondary Outcome: Change From Baseline in the Disease Activity Score 44-Erythrocyte Sedimentation Rate (DAS44-ESR)
Description: Ritchie articular index (RAI); a joint count that grades the tenderness of 26 joints on a scale of 0-3); the number of swollen joints from 44 joints (swollen44); ESR in mm/hour after 1 hour and the patient's global disease activity on a Visual Analogue Scale (VAS) of 100 mm (0=no disease activity to right end of the line 100=maximum disease activity) were used to calculate DAS44-ESR using the following formula: DAS44-ESR = 0.54*sqrt(RAI) + 0.065*(swollen44) + 0.33*ln(ESR) + 0.0072*VAS. Lower numbers were better. A negative change from Baseline indicated improvement.
Time Frame: Baseline and Days 13,27,43,56,71,99 and EOT Up to Day 118
Population: All randomized participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Number analyzed (Participants) | 8 | 7 | 9
score on a scale
  Day 13 (n=8, 7, 9) | -0.473 (0.7412) | -0.310 (0.5369) | -0.344 (0.6491)
  Day 27 (n=8, 7, 9) | -0.798 (0.6432) | -0.995 (0.7094) | -0.383 (0.7425)
  Day 43 (n=8, 7, 8) | -0.873 (0.6064) | -0.852 (0.8223) | -0.469 (0.6585)
  Day 56 (n=8, 6, 8) | -1.002 (0.9624) | -1.190 (0.8217) | -1.184 (1.0178)
  Day 71 (n=7, 6, 7) | -0.853 (0.4461) | -0.980 (0.7478) | -1.134 (1.1240)
  Day 99 (n=8, 6, 8) | -0.678 (0.4345) | -0.914 (0.7782) | -1.025 (0.8533)
  EOT (n=8, 6, 9) | -0.591 (0.5664) | -0.974 (0.5992) | -1.138 (0.9667)

ADVERSE EVENTS:
Time Frame: From Day 1 Up to Day 118
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Namilumab 150 mg | Namilumab 300 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 5/8 | 4/7 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Namilumab 150 mg (N=8) | Namilumab 300 mg (N=7) | Placebo (N=9)
Non-small cell lung cancer stage IIIa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Namilumab 150 mg (N=8) | Namilumab 300 mg (N=7) | Placebo (N=9)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Vitreous detachment (Eye disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 1
Body temperature increased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0
Blood pressure systolic increased (Investigations) | 1 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0
Haemoglobin urine present (Investigations) | 0 | 1 | 0
Mean cell volume increased (Investigations) | 0 | 0 | 1
Red blood cell sedimentation rate increased (Investigations) | 1 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 1 | 0
Urine ketone body present (Investigations) | 0 | 0 | 1
White blood cell count increased (Investigations) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.